CLINICAL TRIAL: NCT01183520
Title: Effect of High Omega-3 Fish Intake on Lipid Peroxidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); University of North Dakota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GFHNRC017
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Omega-3 Fatty Acids; Lipid Peroxidation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 90 grams of Salmon (Active Comparator): Subjects will consume 90 grams of salmon twice a week for 4 weeks
  Interventions: Dietary Supplement: Omega-3 fish oil provided by salmon
- 180 grams of salmon (Active Comparator): Subjects will consume 180 grams of salmon twice a week for 4 weeks
  Interventions: Dietary Supplement: Omega-3 fish oil provided by salmon
- 270 Grams of Salmon (Active Comparator): Subjects will consume 270 grams of salmon twice a week for 4 weeks
  Interventions: Dietary Supplement: Omega-3 fish oil provided by salmon

INTERVENTIONS:
Dietary Supplement: Omega-3 fish oil provided by salmon — Eating 3 different amounts of provided salmon twice a week for four weeks

SUMMARY:
The overall goal of this project is to identify an appropriate level of high omega-3 fish (salmon) consumption that will promote optimal omega 3 nutritional status without increasing the level of lipid oxidation in the body.

DETAILED DESCRIPTION:
Studies have demonstrated that the intakes of fatty fish and fish oils are associated with decreases in cardiovascular disease and other chronic disease states. This is related to the long chain omega-3 fatty acid (n-3) content of fish and fish oil, specifically eicosapentaenoic acid and docosahexaenoic acid. Although the consumption of high n-3 fish is recommended in the 2005 US Dietary Guidelines for Americans, no specific consumption levels are made for the fatty acid eicosapentaenoic acid (EPA) and/or the fatty acid docosahexaenoic acid (DHA) or total fish intake.

Consumption of high n-3 fish or dietary supplementation of fish oil will lead to increased levels of these fatty acids in plasma lipoproteins, cell and tissue lipid. This change in membrane lipid is thought to be responsible for the anti-inflammatory effects of n-3. Because highly unsaturated fatty acid are subject to peroxidation, the level of fish intake that is sufficient to modify membrane n-3 content and the exact level that enhances peroxidation is unknown.

We will perform a dose-response feeling study in which varied levels of fish (salmon) will be provided in random order separated by 4 or more week washout periods. We will assess the level of cell membrane enrichment with n-3 and the effect on lipid peroxidation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-34.9
* Non-smoker
* Free of major medical conditions
* Willing to comply with protocol requirements

Exclusion Criteria:

* Use of lipid modifying drugs or supplements
* Taking fish oil or flax supplements
* Regular fish consumer
* Planning to gain to lose weight
* Pregnant or lactating

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Long chain omega-3 fatty acid (n-3) | 6 months
  Effect of different levels of n-3 intake on n-3 fatty acids in plasma lipoproteins, cell and tissue lipids (cell enrichment)

SECONDARY OUTCOMES:
lipid peroxidation | 6 months
  Effect of different levels of n-3 intake on lipid peroxidation

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Picklo, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA ARS Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Background] Holman RT. Control of polyunsaturated acids in tissue lipids. J Am Coll Nutr. 1986;5(2):183-211. doi: 10.1080/07315724.1986.10720125. PMID 2873160
- [Background] Raatz SK, Bibus D, Thomas W, Kris-Etherton P. Total fat intake modifies plasma fatty acid composition in humans. J Nutr. 2001 Feb;131(2):231-4. doi: 10.1093/jn/131.2.231. PMID 11160538
- [Background] Roberts LJ 2nd, Montine TJ, Markesbery WR, Tapper AR, Hardy P, Chemtob S, Dettbarn WD, Morrow JD. Formation of isoprostane-like compounds (neuroprostanes) in vivo from docosahexaenoic acid. J Biol Chem. 1998 May 29;273(22):13605-12. doi: 10.1074/jbc.273.22.13605. PMID 9593698
- [Background] Song WL, Paschos G, Fries S, Reilly MP, Yu Y, Rokach J, Chang CT, Patel P, Lawson JA, Fitzgerald GA. Novel eicosapentaenoic acid-derived F3-isoprostanes as biomarkers of lipid peroxidation. J Biol Chem. 2009 Aug 28;284(35):23636-43. doi: 10.1074/jbc.M109.024075. Epub 2009 Jun 11. PMID 19520854
- [Background] Roberts LJ 2nd, Fessel JP. The biochemistry of the isoprostane, neuroprostane, and isofuran pathways of lipid peroxidation. Chem Phys Lipids. 2004 Mar;128(1-2):173-86. doi: 10.1016/j.chemphyslip.2003.09.016. PMID 15037162
- [Derived] Raatz SK, Scheett AJ, Johnson LK, Jahns L. Validity of electronic diet recording nutrient estimates compared to dietitian analysis of diet records: randomized controlled trial. J Med Internet Res. 2015 Jan 20;17(1):e21. doi: 10.2196/jmir.3744. PMID 25604640
- See also: USDA Grand Forks Human Nutrition Research Center — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/